CLINICAL TRIAL: NCT03909451
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Ascending Multiple-dose Study to Determine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Orally Administered Sotagliflozin in Healthy Chinese Subjects
Brief Title: Sotagliflozin Multiple-dose Study in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TDR15349; U1111-1199-6171 (Other: UTN)
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 (Experimental): Sotagliflozin dose 1, once daily for 8 days
  Interventions: Drug: Sotagliflozin (SAR439954)
- Dose 2 (Experimental): Sotagliflozin dose 2, once daily for 8 days
  Interventions: Drug: Sotagliflozin (SAR439954)
- Placebo (Placebo Comparator): Placebo, once daily for 8 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Dose 1; Dose 2
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the safety and tolerability of sotagliflozin after a multiple oral dose administration in Chinese healthy subjects.

Secondary Objectives:

* To assess the pharmacokinetic (PK) parameters of sotagliflozin after a multiple oral dose administration in Chinese healthy subjects.
* To assess the pharmacodynamics (PD) parameters of absolute urinary glucose excretion after a multiple oral dose administration in Chinese healthy subjects.

DETAILED DESCRIPTION:
The study duration per subject will be up to 41 days and will consist of a screening period of up to 28 days, a dosing period of 8 days, and a follow up visit 5 days after last dosing.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 45 years of age, inclusive.
* Body weight between 50.0 and 95.0 kg, inclusive, for male or female subjects; body mass index between 18.5 and 27.9 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination), vital signs, electrocardiogram, and clinical laboratory parameters.

Exclusion criteria:

* Any history or presence of clinically relevant illness at screening, which could interfere with the objectives of the study or the safety of the subject's participation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation any volume, within 2 months before inclusion.
* Symptomatic postural hypotension.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* If female, pregnancy, breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 41 days
  Proportion of patients who experienced adverse events/treatment-emergent AEs (TEAE)

SECONDARY OUTCOMES:
Assessment of PK parameter: Maximum plasma concentration (Cmax) | On Day 1 and from Day 8 to Day 13
  Sotagliflozin and Sotagliflozin-O-glucuronide: Maximum plasma concentration (Cmax)
Assessment of PK parameter: Area under curve from 0 to 24 hours (AUCtau) | On Day 1 and Day 8
  Sotagliflozin and Sotagliflozin-O-glucuronide: Area under curve from 0 to 24 hours (AUCtau) of sotagliflozin
Assessment of PK parameter: Area under the concentration-time curve (AUC) | From Day 8 to Day 13
  Sotagliflozin and Sotagliflozin-O-glucuronide: Area under the concentration-time curve from 0 to infinity
Assessment of PD parameter: urinary glucose excretion (UGE) | On Day 1 and Day 8
  Total 24-hour urinary glucose excretion (UGE) after dose with sotagliflozin

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 1560001, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org